CLINICAL TRIAL: NCT03189108
Title: Collection of Malignant Ascites, Pleural Fluid and Blood From Patients With Solid Tumors
Brief Title: Collection of Malignant Ascites, Pleural Fluid, and Blood From People With Solid Tumors
Status: Terminated | Type: Observational
Why Stopped: PI left NIH
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170100; 17-C-0100
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Cancer
Keywords: Malignant Effusion Composition; Paracentesis; Thoracentesis; Natural History
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with a diagnosis of malignant solid tumor

SUMMARY:
Background:

Researchers want to study fluids and blood of people with cancer. The fluids are from the abdomen and around the lungs. Studying these might help researchers learn about the biology of cancer. This may lead to better ways to treat cancer.

Objectives:

To study the biology of cancer.

Eligibility:

Adults 18 and older with malignant solid tumors.

Design:

Participants will be screened with medical history, blood tests, and confirmation of diagnosis.

Participants will have samples taken at regularly scheduled procedures. Fluids from the abdomen and/or lungs will be taken as part of the procedures. Blood will be taken separately.

Participants may be asked to give more samples at future procedures.

DETAILED DESCRIPTION:
Background:

-Malignant ascites or pleural effusions are often seen in patients with solid tumor

malignancies.

-Malignant ascites is proinflammatory with many cytokines present and acts to promote

tumor cell growth.

-The cellular composition of malignant ascites consists of lymphocytes, macrophages and

monocytes.

-Serum monocytes and lymphocytes play a role in the native host anti-tumor immune

mediated mechanisms.

-A paracentesis or thoracentesis is often done for symptomatic relief from the malignant

fluid collection.

Primary Objective:

-To obtain blood samples and ascites and pleural effusion samples from patients with solid

tumor malignancies, with the intent of performing translational studies related to cancer.

Eligibility:

* Patients greater than or equal to 18 years of age.
* Diagnosis of malignant solid tumor.
* Patients must be able and willing to provide informed consent.

Design:

-We will collect approximately 200cc-5L ascites from patients that are undergoing a

therapeutic paracentesis or thoracentesis. No thoracentesis or paracentesis will be

performed solely for research purposes.

-The fluid will be collected during the medical procedure and may be collected at more

than one time point.

-We will also collect 30ml of peripheral blood. This will be from patients who are being

seen in follow up, consultation, or presenting for enrollment on a clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants greater than or equal to 18 years of age with histologically proven malignant solid tumors
* Ability and willingness to provide informed consent to participation.
* Participants with malignant solid tumors with a clinical indication for a thoracentesis or paracentesis.

EXCLUSION CRITERIA:

-Children < 18 years of age are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being seen in follow up, consultation, or presenting for enrollment on a clinical trial at the NIH Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
To obtain blood samples, ascites and pleural effusion samples from patients with solid tumor malignancies, with the intent of performing translational studies related to cancer. | Ongoing
  Experimental - Translational study outcomes from the collection/analysis of blood samples; and ascites and pleural effusion samples from patients with solid tumor malignancies.

SECONDARY OUTCOMES:
Develop the malignant fluid as a culture model to replicate intraperitoneal growth of ovarian cancers. | ongoing
Characterize malignant effusion composition through immunohistochemistry and flow cytometry. | ongoing
Compare immune cell phenotype in ascites and blood from the patient. | ongoing
Study in vivo characteristics of matched tumor cells and peripheral blood leukocytes from the same patient in xenograft models | ongoing
Establish a bank of clinically annotated samples for translational science. | ongoing
Compare selected matched sets of samples from the same patient to evaluate both for treatment response. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0100.html